CLINICAL TRIAL: NCT07309835
Title: Capturing Ethnic Minority Experiences of Genomic Pathways to Understand What Changes Are Needed to Promote Greater Equity Within the Genomic Medicine Service.
Brief Title: Improving Genetic Medicine for Ethnic Minority Groups
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 360821
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Genetic Testing
Keywords: interview; ethnic minority; mixed method; qualitative; genetic testing; genomic testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lay members of the public: Lay members of the public recruited from community settings
- Community organisers and charity workers: Community and charity workers recruited from community settings
- Patients, family members and carers: Recruited through a mixture of healthcare and community settings
- Healthcare professionals: Recruited through professional networks

SUMMARY:
A key aim of the nationally commissioned Genomic Medicine Service (GMS) in England is to encourage equity of access between different patient groups, however, there is evidence to suggest that it is being under-utilised by ethnic minority groups. The aim of this study is to explore how ethnic minority populations interact with the GMS and to identify changes that would promote equity within those services.

This is a mixed-methods study using interviews and group discussions with lay people, community organisers and charity workers, people who have had direct or indirect contact with the genomic medicine service and professionals within the service. By including potential service users, service users and professionals in this work and allowing people to share their experiences in whatever method feels most comfortable to them, we aim to get a broad understanding of the lived experience of everyone involved in these pathways which will be key to gaining a holistic understanding of how they are working in real world settings.

The primary outcome measure will be an increased understanding of the experiences of people from ethnic minority groups navigating the genomic medicine space. The secondary outcome measure will be an increased understanding of how experiences differ across and between ethnic groups. We intend to use our insights to recommend structural changes which will improve utilisation of the genomic medicine service by patients from ethnic minority groups.

DETAILED DESCRIPTION:
In 2019 a nationally commissioned Genomic Medicine Service (GMS) was established to deliver high-quality genomic testing for patients affected by rare diseases and cancer in England. A key aim of the new GMS was to encourage equity of access between different patient groups, including ethnic minority groups. A report produced by the NHS Race and Health Observatory in 2024 pointed to several barriers which remain to be addressed in trying to ensure that people from diverse backgrounds can access GMS services and genomic research and highlighted that a paucity of ethnicity recording makes it difficult to measure equity of access between different ethnic groups.

Insights into the lived experiences of ethnic minority groups with reference to genomic testing in the UK are limited. Even when studies have included diverse voices, they are often aggregated with other minority ethnic groups, assuming collective experiences.

We will conduct interviews and group discussions with lay people, community organisers and charity workers, people who have had direct or indirect contact with the genomic medicine service and professionals within the service. Some of our participants will be recruited from community settings. Others will be recruited from healthcare settings where they will be identified from a mixture of retrospective and prospective recruitment.

The overarching aim of this study is to capture the experiences of ethnic minority populations within regional genomic medicine services and to identify specific changes that are needed to promote equity and cultural competence within those services. While we recognise that it will not be possible to derive recommendations which are applicable across all ethnic minority groups and the entire GMS, our work will serve as an exemplar to others who wish to undertake similar work with their specific population.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Have capacity to consent to take part

Exclusion Criteria:

* Under 18 years of age
* Affected by a serious mental health condition
* Learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is individuals who identify as being from ethnic minority backgrounds and community organisers, charity workers and health care professional who have insight into their experiences
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2031-01-30 (Estimated); Study Completion 2031-01-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative insights into people's experiences | 5 years
  increased understanding of the experiences of people from ethnic minority groups navigating the genomic medicine space

SECONDARY OUTCOMES:
Qualitative insights into differences between minority groups | 5 years
  increased understanding of the experiences of people from ethnic minority groups navigating the genomic medicine space

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas' NHS foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The protocol will be shared. No personal identifiers will be shared with other researchers, but de-identified transcripts will be shared on application to the CI.
Supporting Information: Study Protocol
Time Frame: For 2 years after the end of the study.
Access Criteria: On application to the CI.